CLINICAL TRIAL: NCT06398743
Title: CORRECT-MRD I: First Colorectal Cancer Clinical Validation Study to Predict Recurrence Using a Circulating Tumor DNA Assay to Detect Minimal Residual Disease
Brief Title: First CORRECT Study of Minimal Residual Disease (MRD) Detection in Colorectal Cancer
Acronym: MRD
Status: Active, not recruiting | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-001
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal; ctDNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Stage II or III: Patients with stage II or III colorectal cancer
  Interventions: Device: MRD

INTERVENTIONS:
Device: MRD — ctDNA MRD test

SUMMARY:
The CORRECT - MRD I study will prospectively enroll patients who have undergone complete surgical resection for stage II or III colorectal cancer. Patients will be followed for up to 5 years for recurrence.

ELIGIBILITY:
Inclusion Criteria:

Subject is/has:

1. 18 years of age or older.
2. Diagnosis of carcinoma of the colon or rectum (patients with lymphomatous, sarcomatous,or neuroendocrine features are not eligible).
3. Post complete surgical resection of CRC, with last surgery occurring within 180 days prior to enrollment are eligible if all of the following conditions are met:

   1. in the opinion of the surgeon, all grossly visible tumor was completely resected ("curative resection") and
   2. histologic evaluation by the pathologist confirms the margins of the resected specimens are not involved by malignant cells.

   i. Patients with T4 tumors that have involved an adjacent structure (e.g., bladder, small intestine, ovary, etc.) by direct extension form the primary tumor must have had all or a portion of the adjacent structure removed en bloc with the primary tumor and local radiation therapy will not be utilized.
4. Pathologic Stage II or III CRC.
5. ECOG performance status ≤ 2 (0, 1 or 2).
6. Able to understand and provide written informed consent.
7. Willing and able to comply with the study requirements, which includes the collection of approximately 35mL of blood for each research blood draw.

Exclusion Criteria:

Subject is/has:

1. Initiated adjuvant therapy for current CRC diagnosis (note: neoadjuvant therapy acceptable).
2. Known pregnancy or breastfeeding at time of enrollment.
3. Prior history of any invasive cancer (including CRC) within the past 3 years prior to informed consent, with the exception of non-melanoma skin cancer. Patients with a prior history of noninvasive (in situ) carcinomas may participate after definitive treatment.
4. Prior transplant history:

   1. Prior allogeneic hematopoietic stem cell transplant at any time.
   2. Prior solid organ transplant within the last 2 years prior to enrollment.
5. Multiple cancer diagnoses: Synchronous or asynchronous diagnoses (or suspicion) of multiple primary cancers at the time of eligibility screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who have undergone surgery for stage II or III colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To validate the association of post-definitive therapy and pre-recurrence follow-up ctDNA positivity with Recurrence Free Interval, defined as elapsed time from surgical resection to the first clinical recurrence or CRC-related death. | 6 years

SECONDARY OUTCOMES:
Time from the first ctDNA positivity to recurrence among subjects who have a positive ctDNA finding and have recurred. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Somasundaram Subramaniam, MD, Study Director — Exact Sciences
Locations (22):
- Israel (6):
  - Tel Aviv Sourasky Medical Center, Tel Aviv Yaffo, Central District
  - Hillel Yaffe Medical Center, Hadera, North
  - Soroka University Medical Center, Beersheba, Southern District
  - HaEmek Medical Center, Afula
  - Hadassah University Hospital - Mount Scopus, Jerusalem
  - Shaare Zedek Medical Center Jerusalem, Jerusalem
- Italy (3):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale Tumori - Fondazione G Pascale, Napoli
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kagawa University Hospital, Kita-gun
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncológico Clara Campal (HM CIOCC), Madrid
- United Kingdom (8):
  - Churchill Hospital, Headington, Oxford
  - Edinburgh Cancer Centre, Edinburgh, Scotland
  - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Worcestershire Royal Hospital, Worcester, Worcestershire
  - Ipswich Hospital, Ipswich
  - Kidderminster Hospital and Treatment Centre, Kidderminster
  - Alexandra Hospital, Redditch
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include test, tables, figured, and appendices. The study protocol, statistical analysis plan (when applicable), informed consent form (when applicable). May not be reproduced nor disseminated outside of Exact Sciences without permission and the clinical study report (when applicable) will also be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from 2 years and ending 4 years after publication
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary institutional review board/independent ethics committee approvals or waivers as applicable to conduct research.